CLINICAL TRIAL: NCT01566500
Title: Best Practices and Challenges in Medication Adherence for Individuals With Epilepsy
Brief Title: Medication Adherence in Individuals With Epilepsy
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Epilepsy Foundation (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Niall Bolger, Professor of Psychology, Columbia University
Other Study IDs: AAAI1597
Record Dates: First submitted 2012-03-28; First posted 2012-03-29 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Medication Adherence
MeSH Terms: conditions — Epilepsy; Medication Adherence

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is an urgent need to understand the psychological and situational factors that influence medication adherence in individuals with epilepsy. According to the Center for Disease Control (CDC, 2010) about 2.5 million people in the United States have epilepsy and one third of them still have seizures despite receiving treatment. With proper medication, an estimated 60-70% of individuals with new onset epilepsy become, and remain, seizure free (Kwan & Brodie, 2000). Despite the success of medical treatment of epilepsy, many patients do not receive these benefits due to inadequate adherence to medication (Meyer et al., 2010). And, as with other chronic medical conditions, estimates suggest that between 30% and 60% of patients with epilepsy are not adherent with their drug regimens (Green & Simons Morton, 1988; Leppik, 1990; Jones et al., 2006). Poor adherence may be the most important cause of poorly controlled epilepsy (Gomes et al., 1998). Stanaway et al. (1985) found that 31% of seizures were precipitated by nonadherence to medication.

Questions regarding adherence are theoretically informed by Fisher et al. (2006)'s Information Motivation Behavioral Skills (IMB) model. While originally developed to describe, predict, and inform interventions for antiretroviral treatment for human immunodeficiency virus (HIV), this study applies the model to epilepsy for the first time. In addition, this study intends to produce an accurate description of how individuals with epilepsy manage their medication adherence by identifying current self regulation strategies (immediate adherence behaviors, preparatory behaviors, and barrier management strategies) and their situational determinants. Situational determinants can explain some of the fluctuations in medication adherence. Patients who are motivated to take their medications might still show inconsistent medication adherence. For example, patients might miss good opportunities to take their medication or fail to anticipate unexpected barriers such as a spontaneous dinner with friends or a bout of depression. Therefore, the study will take particular care to investigate situational cues such as good opportunities for adherence (e.g., taking medication with regular meals or before brushing teeth) and expected and unexpected barriers. Preparatory behaviors and their cues are also of interest in this study: Some patients use facilitators (such as physical or electronic reminder systems, electronic pill bottles and pill boxes) to ensure adequate medication adherence. Social support can serve a similar function of reminding patients to take their medication. To address these questions, the investigators plan to explore how individual regulation and social support influence medication adherence in patients with epilepsy. The specific aims of the proposed research are:

1. To test the hypothesis that there will be a main effect of information, motivation and behavioral skills, on adherence behavior, and that a mediation model will show that information and motivation effects are partially mediated through behavioral skills.
2. To identify self regulation strategies and their situational cues (good opportunities, facilitators, and barriers) for medication adherence among individuals with epilepsy to better describe best practices and challenges.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Epilepsy

Exclusion Criteria:

* Age (under 18, over 65)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 140 participants between 18 and 65 years old will be recruited with the condition that all participants have been diagnosed with epilepsy. The participants will be of diverse ethnic background. It is estimated that the participant population will also include individuals from a disadvantaged socioeconomic and/or educational background.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niall Bolger, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Morningside Campus, New York, New York, United States

REFERENCES:
- [Derived] Chesaniuk M, Choi H, Wicks P, Stadler G. Perceived stigma and adherence in epilepsy: evidence for a link and mediating processes. Epilepsy Behav. 2014 Dec;41:227-31. doi: 10.1016/j.yebeh.2014.10.004. Epub 2014 Nov 1. PMID 25461221

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Sample: Adults with self-reported epilepsy.
Period: Overall Study
Arm/Group | Study Sample
Started | 140
Completed | 140
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults with self-reported epilepsy.
Arm/Group | Study Sample
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.51 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 140

OUTCOME MEASURES:

1. Primary Outcome: Raw Count of Number of Days of Medication Nonadherence
Description: The primary outcome of this study is medication adherence as measured by self report with a 4 day recall adherence questionnaire (Chesney, Ickovics, Chambers, et al., 2000).
  The total number of Nonadherence days were counted, then divided by the total number of days for all participants.
Time Frame: Enrollment
Population: Adults with self-reported epilepsy.
Measure: Number; unit: % of nonadherence days
Arm/Group | Study Sample
Number analyzed (Participants) | 140
% of nonadherence days | 28

2. Secondary Outcome: Score on Barriers to Medication Adherence
Description: The Chesney Adherence Questionnaire will be used to measure side effects, drug use and other barriers to medication adherence. The items pertaining to barriers to medication adherence were assessed the same day as enrollment and have a four-week recall period.
Time Frame: Enrollment
Reporting Status: Not Posted

3. Secondary Outcome: Score of Psychosocial Predictors of Adherence
Description: The Fisher IMB (Information-Seeking, Motivation and Behavior) adherence questionnaire will measure what psychosocial factors that act as predictive of medication adherence. The items pertaining to barriers to medication adherence were assessed the same day as enrollment and have a twelve month recall period.
Time Frame: Enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: It was an observational study where none of the participants were at risk during the study hence the meaning of "0" Total Number of Participants at Risk.
Arm/Group | Study Sample
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No